CLINICAL TRIAL: NCT05813457
Title: Impact of an Early Identification Program for First-Episode Psychosis on the Duration of Untreated Psychosis. Multicenter, Randomized Stepped-wedge Study
Brief Title: Impact of an Early Identification Program for First-Episode Psychosis on the Duration of Untreated Psychosis
Acronym: PRESTO
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 19PH228; 2021-A00787-34 (Other: ANSM)
Record Dates: First submitted 2023-04-03; First posted 2023-04-14 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Psychotic Episode
Keywords: Schizophrenia; Psychiatric centers; psychiatric illnesses; psychiatric care
MeSH Terms: conditions — Schizophrenia; Mental Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PRESTO program (Experimental): The PRESTO programs consists of an early identification program for First Episod Psychosis, called PRESTO (First Episodes Raise Awareness Treat Referral), including 3 complementary components:
  * Information campaign for the general population
  * Training of front-line actors
  * Facilitating access to specialized care by setting up mobile teams made up of "pivotal" workers who provide the link between front-line actors and specialized psychiatric care
  Interventions: Other: PRESTO Early Identification Program
- Usual Care (No Intervention): No change in the conditions of referral of First Episod Psychosis (emergencies, hospitalizations, consultations)

INTERVENTIONS:
Other: PRESTO Early Identification Program — The program combines :
  1. A population-based information component (information campaign aimed at the general population).
  2. A training component for the LPAs (Front Line Actors: general practitioners, school and university medicine, pharmacists, teenagers school and university medicine, pharmacists, teenagers' homes, association networks, SAMU, firemen, etc.).
  3. Facilitated access to care for FPE patients in the form of a "pivot" mobile team that can directly meet the patient at the request of the LPA, initiate care and ensure the relay within a the relay within 4 weeks to the existing specialized psychiatric structures on the site (CMP, CATTP (CMP, CATTP, day hospital, hospitalization unit, child and adolescent psychiatry services) adolescent psychiatry services)
  Other Names: PRESTO Program
  Arms: PRESTO program

SUMMARY:
The First-Episode Psychosis (FPE) is a severe disorder that can include delusions, cognitive disorders and suicidal behavior. In the majority of cases (more than 80%) it evolves into schizophrenia. Numerous studies show that the rapidity of the initial management of FPE would reduce the risk of negative evolution and would have a decisive impact on the short and long term prognosis. The rapidity of this management can be measured by the duration of untreated psychosis, or DUP (Duration of Untreated Psychosis), the time interval between the appearance of the first frank psychotic symptoms and the initiation of adequate psychiatric care. The objective of this study is to show the impact of an intervention facilitating access to specialized care for PEP on the reduction of DUP. This intervention consists of an early identification program for FPE, the PRESTO program, specifically targeting 3 determining steps in the reduction of DUP:

* Informing the general population about psychotic disorders
* Knowledge of front line actors (APL: general practitioners, school and university medicine, teenager's house, associative networks educators, emergency services, firefighters, etc.) about FPE and its management
* Articulation between APL and specialized psychiatric care

DETAILED DESCRIPTION:
The DUP is an easily measurable indicator, closely linked to prognosis and potentially modifiable, which has led to its wide use to guide the development of early identification programs. Great disparities exist across the world, between different countries and even different regions. France is unusually late, with an average DUP of at least 18 months. Several elements may contribute to explain this state in France: absence of a specific care program for FPE in the vast majority of psychiatric centers, significant stigmatization of psychiatric illnesses, the opacity of psychiatric care and of psychiatric care and lack of knowledge of its organization, in particular by the primary care network that receives patients with PEP in the first line. To date, there is no systematic program in France designed to rapidly identify FPE patients and hasten their specialized care. The objective of this study is to show the impact of an intervention facilitating access to specialized care for PEP on the reduction of DUP.

In addition, this study will seek to analyze the implementation factors of such an intervention in view of a possible generalization and perpetuation.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a diagnosis of schizophrenia, schizoaffective disorder, schizophreniform disorder, or brief psychotic disorder established according to DMS 5
* Never having taken neuroleptic treatment for antipsychotic purposes, except for the current episode and for a duration of < 6 month
* Oral consent of the patient or, for minors, of his/her parents to participate in the study

Exclusion Criteria:

* Patients already treated and followed for FPE
* Brief psychotic state not requiring specific management

Ages: 15 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 416 (Estimated)
Dates: Start 2023-06-06 (Actual); Primary Completion 2027-02 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Duration of untreated psychosis (DUP) | Baseline
  Defines the time interval between the onset of the first frank psychotic signs noted by the patient and his or her entourage and treatment in specialized psychiatric care

SECONDARY OUTCOMES:
Number of patients still in care | Week 4
  measurement of the number of patients continuing care
Engagement in care | Week 4
  Measurement of engagement in care through the Service Engagement Scale. It is a 14-item questionnaire, scored from 0 to 3, divided into four categories: availability, cooperation, help-seeking attitude and therapeutic adherence. The questionnaire is completed by the clinician.
treatment adherence | Week 4
  Medication Adherence Rating Scale (MARS) is a 10-item self-reporting multidimensional instrument describing three dimensions: medication adherence behavior (items 1-4), attitude toward taking medication (items 5-8) and negative side effects and attitudes to psychotropic medication (items 9-10). The total score ranges from 0-10 with a higher score indicating better adherence.
therapeutic alliance | Week 4
  measurement of the therapeutic alliance with the "Working Alliance Inventory" self-questionnaire given to the patient and the clinician. It is a self-administered questionnaire with a 36-item therapist or caregiver component and a 36-item patient component. Each item is rated from 1 to 7 (never to always). The score range is 36 to 252. Higher score reflect a more positive rating of working alliance.
Customer satisfaction | Week 4
  Measurement of Customer satisfaction by self-questionnaire with 8 items applicable to a population with psychotic disorders. The CSQ-8 scores range from 8 to 32, with higher values indicating higher satisfaction.
Caregiver Burden | Baseline and week 4
  Measurement of Caregiver Burden by the Zarit Burden Interview in Caregivers of Patients is a self-questionnaire given to the caregiver. This questionnaire consists of 22 items rated on a 5-point Likert scale that ranges from 0 (never) to 4 (nearly always) with the sum of scores ranging between 0 to 88. Higher scores indicate greater burden. A score of 17 or more was considered high burden.
Assessment of the context | before the start and after the end of the PRESTO program
  Semi-structured interview wera done with stakeholders of PRESTO program to assess contextual factors that increase or limit the effect of the intervention, integration of the intervention into the care organization scheme, collaboration with inpatient, outpatient and non-healthcare sectors, means identified to sustain the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Eric FAKRA, MD PhD, Principal Investigator — CHU SAINT-ETIENNE
Locations (6):
- France (6):
  - Hospices Civils de Lyon, Bron
  - Chu Clermont-Ferrand, Clermont-Ferrand
  - Chu Grenoble, Grenoble
  - CHU de Montpellier, Montpellier
  - CHU de Nîmes, Nîmes
  - Chu Saint Etienne, Saint-Etienne

IPD SHARING:
Plan to Share IPD: No